CLINICAL TRIAL: NCT00396188
Title: Corneal Analysis - Pathology Detection Aid
Brief Title: Screening Aid to Identify Corneas That May Have Pathologies or Other Conditions
Status: Completed | Type: Observational
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Atlas II-2006-1-v1
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Corneal Diseases
Keywords: Keratoconus; LASIK; Orthokeratology; Pellucid Marginal Degeneration; Refractive Surgery; normal cornea; post myopic LASIK; post hyperopic LASIK; corneal pathologies (e.g. pellucid marginal degeneration)
MeSH Terms: conditions — Corneal Diseases; Keratoconus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Normals: 1. Patients seeking initial laser vision correction that were screened to be good candidates for the procedure.
  2. No history of refractive or other ocular surgery.
  3. No corneal pathologies.
  4. Normal corneal topography.
  5. Contact lens wearers should discontinue use at least 2 weeks for hard contacts, and 3 days for soft lenses prior to imaging.
- Keratoconus: 1. An irregular cornea determined by distorted keratometry mires, distortion of the retinoscopic, or ophthalmoscopic red reflex (or a combination of these)
  2. At least one of the following biomicroscopic signs: Vogt's striae, Fleischer's ring of >2 mm arc, or corneal scarring consistent with keratoconus.
  3. Contact lens wearers should discontinue use preferably 1 day or at least half an hour prior to imaging.
- Myopic Laser Vision Correction: Patients who have undergone myopic:
  1. LASIK
  2. PRK
  3. LASEK
- Hyperopic Laser Vision Correction: Patients who have undergone hyperopic:
  1. LASIK
  2. PRK
  3. LASEK
- Orthokeratology: 1. Patients using specially designed rigid contact lenses to reshape the cornea to temporarily reduce or eliminate refractive error.
- Others: 1. Corneal conditions (diseases/ pathologies/surgeries) that can potentially affect the corneal surface that are not listed above (e.g. pellucid marginal degeneration; postoperative corneal transplant, intra-corneal ring segments, refractive keratotomy, conductive keratoplasty; peripheral ulcerative keratitis, Terrien's marginal degeneration; etc.).

SUMMARY:
The purpose of this study is to determine the ability of a proprietary software screening tool to discriminate normal corneas (front surface of the eye) from previously diagnosed corneal conditions (diseases/surgeries/pathologies) and to determine the repeatabiltity and reproducibility of the Atlas II corneal topographer in normal human corneas.

DETAILED DESCRIPTION:
1. To establish reference values for SF, CIM, and TKM in subjects with normal corneas.
2. To establish reference values for SF, CIM, and TKM in subjects who underwent myopic laser vision correction.
3. To establish reference values for SF, CIM, and TKM in subjects who underwent hyperopic laser vision correction.
4. To establish reference values for SF, CIM, and TKM in subjects who were diagnosed to have keratoconus.
5. To establish reference values for SF, CIM, and TKM in subjects with history of orthokeratology.
6. To establish reference values for SF, CIM, and TKM in subjects with previously diagnosed corneal conditions (diseases/pathologies/surgeries) affecting the corneal surface that are not listed above.
7. To determine the repeatabiltity and reproducibility of the Atlas II corneal topographer in normal human corneas using true elevation data and axial curvature.
8. To determine the sensitivity, specificity, and accuracy of the Pathfinder II Corneal Analysis software in discriminating normal corneas from previously diagnosed corneal conditions (diseases/pathologies/surgeries) affecting the corneal surface (Phase II).

ELIGIBILITY:
Inclusion Criteria:

Normals

* Patients seeking initial laser vision correction that were screened to be good candidates for the procedure.
* No history of refractive or other ocular surgery.
* No corneal pathologies.
* Normal corneal topography.
* Contact lens wearers should discontinue use at least 2 weeks for hard contacts, and 3 days for soft lenses prior to imaging.

Keratoconus

* An irregular cornea determined by distorted keratometry mires, distortion of the retinoscopic, or ophthalmoscopic red reflex (or a combination of these)
* At least one of the following biomicroscopic signs: Vogt's striae, Fleischer's ring of >2 mm arc, or corneal scarring consistent with keratoconus.
* Contact lens wearers should discontinue use preferably 1 day or at least half an hour prior to imaging.

Myopic Laser Vision Correction

Patients who have undergone myopic:

* LASIK
* PRK
* LASEK

Hyperopic Laser Vision Correction

Patients who have undergone hyperopic:

* LASIK
* PRK
* LASEK

Orthokeratology

* Patients using specially designed rigid contact lenses to reshape the cornea to temporarily reduce or eliminate refractive error.
* Subjects must be 18 years of age or older; able and willing to make the required visit; and able and willing to give consent.

Exclusion Criteria:

* Patients that underwent corneal transplantation or any ocular surgery for the following categories: normal, keratoconus, and orthokeratology)
* Any active infection or inflammation of the cornea.
* PI decides that subject is not suitable due to medical risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will consist of patients seeking consult in the Principal Investigator's (PI) clinical practice and volunteers responding to the study's advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 769 (Actual)
Dates: Start 2007-02; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Reference values of normal and previously diagnosed corneal conditions by Atlas II corneal topographer | 1-2 hours

SECONDARY OUTCOMES:
Repeatabiltity and reproducibility of the Atlas II corneal topographer in human corneas | 1-2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jon Dishler, M. D., Principal Investigator — Dishler Laser Institute; David J Schanzlin, M. D., Principal Investigator — Shiley Eye Center-University of California San Diego; Dennis Burger, O. D., Principal Investigator — Kaiser Permanente, Oakland; Patrick Caroline, COT, Principal Investigator — Pacific University; Tyson Brunstetter, O. D., Principal Investigator — Naval Training Center-Refractive Surgery Clinic; Kevin Reeder, O.D., Principal Investigator — Carmel Mountain Vision Care Center
Locations (4):
- United States (4):
  - Shiley Eye Center-University of California San Diego, La Jolla, California
  - Carmel Mountain Vision Care Center, San Diego, California
  - Dishler Laser Institute, Greenwood Village, Colorado
  - Pacific University, Forest Grove, Oregon

REFERENCES:
- [Background] Zadnik K, Barr JT, Edrington TB, Everett DF, Jameson M, McMahon TT, Shin JA, Sterling JL, Wagner H, Gordon MO. Baseline findings in the Collaborative Longitudinal Evaluation of Keratoconus (CLEK) Study. Invest Ophthalmol Vis Sci. 1998 Dec;39(13):2537-46. PMID 9856763
- [Background] Twa MD, Parthasarathy S, Roberts C, Mahmoud AM, Raasch TW, Bullimore MA. Automated decision tree classification of corneal shape. Optom Vis Sci. 2005 Dec;82(12):1038-46. doi: 10.1097/01.opx.0000192350.01045.6f. PMID 16357645